CLINICAL TRIAL: NCT02540720
Title: The Research of Standard Diagnosis and Treatment for Severe Henoch-Schonlein Purpura in Children
Brief Title: The Research of Standard Diagnosis and Treatment for Severe HSP in Children
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Children's Hospital (Other)
Responsible Party: Principal Investigator, Aihua Zhang, Hospital vice president, Nanjing Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Zhai
Record Dates: First submitted 2015-08-20; First posted 2015-09-04 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Henoch-Schoenlein Purpura
MeSH Terms: conditions — IgA Vasculitis | interventions — Dexamethasone; gamma-Globulins; Hemoperfusion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- group 1 (Experimental): Dexamethasone 0.5mg/kg.d i.v.
  Interventions: Drug: Dexamethasone
- group 2 (Experimental): Dexamethasone & gamma globulin Dexamethasone 0.5mg/kg.d i.v. & gamma globulin i.v. qd*3d, and the total dose is 2g/kg
  Interventions: Drug: Dexamethasone; Drug: Gamma globulin
- group 3 (Experimental): Dexamethasone & hemoperfusion Dexamethasone 0.5mg/kg.d i.v & hemoperfusion should be given at least three times in five days
  Interventions: Drug: Dexamethasone; Procedure: Hemoperfusion

INTERVENTIONS:
Drug: Dexamethasone
Drug: Gamma globulin
  Arms: group 2
Procedure: Hemoperfusion
  Arms: group 3

SUMMARY:
This study is performed to evaluate the efficacy and safety of various measures in the treatment of severe HSP in children.

DETAILED DESCRIPTION:
Henoch-Schonlein purpura (HSP) is a systemic vasculitis affecting small vessels with immunoglobulin A (IgA)-dominant immune deposits. The clinical manifestations of severe HSP vary from massive hemorrhage and necrosis of the skin to severe gastrointestinal symptoms. The course of the disease would encounter delay and relapse. To some extent, the traditional therapy alleviate the clinical symptoms, but fail to timely clear up the immune depositions, causing the damage to the kidney.

In the study, the patients will be given dexamethasone 0.5mg/kg/d, then be randomised to receive either gamma globulin i.v. or hemoperfusion if the disease can't be controlled with steroid treatment for more than two days.

The investigators will explore the biological markers and compare the efficacy and safety of both measures in the treatment of serve HSP in children. The purpose of the study is to optimize the treatment of severe HSP for children with different ages.

ELIGIBILITY:
Inclusion Criteria:

* Severe HSP: could not be controlled with dexamethasone 0.5mg/kg/d or the total dose above 20mg/d for more than two days

Exclusion Criteria:

* The children with congenital diseases

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2015-08; Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
The Symptoms of Digestive Tract | 2 weeks
  The stomachache and other symptoms of digestive tract disappear
The Symptoms of Joint System | 2 weeks
  The arthralgia disappears

SECONDARY OUTCOMES:
The Skin Rash | 2 weeks
  The Skin Rash disappears
Renal function | 2 weeks
  There is no damage in kidney.

CONTACTS AND LOCATIONS:
Overall Officials: Aihua Zhang, M.D., Study Chair — Department of Nephrology, Nanjing children's hospital
Locations (1):
- Nanjing Children's Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Hahn D, Hodson EM, Craig JC. Interventions for preventing and treating kidney disease in IgA vasculitis. Cochrane Database Syst Rev. 2023 Feb 28;2(2):CD005128. doi: 10.1002/14651858.CD005128.pub4. PMID 36853224